CLINICAL TRIAL: NCT06221085
Title: The Influence of Body Mass Index and Smartphone Overuse on Cervical Myofascial Pain in College-aged Female Students: A Cross-sectional Study
Brief Title: The Influence of Body Mass Index and Smartphone Overuse on Cervical Myofascial Pain: A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Wafaa Mahmoud Amin, Lecturer, University of Jazan
Other Study IDs: HAPO-10-Z-003
Record Dates: First submitted 2024-01-13; First posted 2024-01-24 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Cervical Myofascial Pain Syndrome; Smartphone Addiction; Body Weight; Obesity
MeSH Terms: conditions — Internet Addiction Disorder; Body Weight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal BMI: 30 female students who have normal BMI <25kg/m2.
  Interventions: Diagnostic Test: Pain Pressure Threshold (PPT)
- overweight: 30 female students who are overweight and their BMI 25 - 30 kg/m2
  Interventions: Diagnostic Test: Pain Pressure Threshold (PPT)
- obese: 30 female students who are obese and their BMI > 30 kg/m2.
  Interventions: Diagnostic Test: Pain Pressure Threshold (PPT)

INTERVENTIONS:
Diagnostic Test: Pain Pressure Threshold (PPT) — Researchers measure pain pressure thresholds (PPTs) by applying a Pressure gauge algometer (PGA) over the myofascial trigger points (TrPs) on the body. PPT is defined as the lowest stimulus intensity at which a subject perceives pain.
  The clinician applies it perpendicular to the long axis of the structure on which it is placed. The examiner increases the pressure at a rate of 1 kg/s until the subject feels pain or discomfort, and then the PPT values are measured three times for each muscle. Participants verbally report the first sensation of pain or discomfort, at which point the examiner stops the pressure.
  Other Names: PPTs

SUMMARY:
An observational cross-sectional study will be conducted on 90 female students (right dominant) aged 19-26 years at Jazan University, they will have 40 points or more on Smartphone Addiction Proneness Scale (SAPS) and will be divided into three groups (30 students for each): Group I (BMI<25kg/m2), Group II (BMI 25-30kg/m2), and Group III (BMI >30 kg/m2). Pain pressure thresholds were measured using a pressure gauge algometer (PGA) over trigger points in the neck muscles.

DETAILED DESCRIPTION:
Materials and Methods

Study design:

This is an observational cross-sectional design will be conducted on female subjects from Applied Medical College, Jazan University, Kingdome of Saudi Arabia.

Participants:

A study will be conducted on 90 female students from Jazan University based on the following:

The study will be conducted according to the tenets of the Declaration of Helsinki, and registered in the clinical registry after getting the ethical approval from the Standing Committee for Scientific Research at Jazan University. The sample size is determined using G-Power software (Universities, Düsseldorf, Germany) with a power of 80%, a p-value of 0.05, and an effect size of 0.5. A sample size of 75 (25 individuals in each group) individuals will be included in the study, and to compensate for the dropout rate, the sample size will be increased by 20% in each group to be 30 individuals in each group. The Participants will be divided according to the BMI into three groups: Group I: 30 female students who have normal BMI <25kg/m2. Group II: 30 female students who are overweight and their BMI 25 - 30 kg/m2. Group III: 30 female students who are obese and their BMI > 30 kg/m2.

Measurements:

Body mass index assessment and calculation:

Investigators will measure the height of the participants using a stadiometer with a calibrated analog scale and the weight using a Breuer electronic scale with an accuracy of 0.01 kg.

Pain Pressure Threshold (PPT):

The examiner identifies a trigger point by palpating and applying vertical pressure to the skin. Once identified, the clinician guides the tip of Pressure gauge algometer (PGA) between the finger and thumb to avoid slipping along rounded contours. The clinician applies it perpendicular to the long axis of the structure on which it is placed. The examiner increases the pressure at a rate of 1 kg/s until the subject feels pain or discomfort, and then the PPT values are measured three times for each muscle. Participants verbally report the first sensation of pain or discomfort, at which point the examiner stops the pressure.

PPT of upper fiber of trapezius muscle: The upper trapezius trigger point is located in the more horizontal fibers of the upper trapezius at the back of the shoulder, about halfway between the spine and the acromion.

Sternocleidomastoid (SCM) PPT:

TrPs are in the upper part of the sternal division of the muscle, near its insertion into the mastoid process. TrPs are in the middle part of this division. TrPs are at the lower end of this division, near its attachment to the sternum.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 26 years.
* Participants who send at least 25 text messages or emails per day.
* Use their smartphone to browse the Internet, and/or play games for more than one hour per day.
* If participants score on the Smartphone Addiction Scale (SAPS) > 40 points.
* Right dominant hand.

Exclusion Criteria:

Any subject will be excluded from the study if they meet one or more of the following criteria:

* Neck musculoskeletal trauma.
* Congenital deformities.
* Surgical or neurological disease.
* History of neck injury, and pregnancy.

Ages: 19 Years to 26 Years | Sex: Female
Age Groups: Adult
Study Population: A study will be conducted on 90 female students from Jazan University
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
PPT of upper fiber of trapezius muscle | two minutes
  The upper trapezius trigger point is located in the more horizontal fibers of the upper trapezius at the back of the shoulder, about halfway between the spine and the acromion.

SECONDARY OUTCOMES:
PPT of Upper Part of Sternocleidomastoid (SCM) | two minutes
  TrPs are in the upper part of the sternal division of the muscle near its insertion into the mastoid process.
PPT of middle Part of Sternocleidomastoid (SCM) | two minutes
  TrPs are in the middle part of this division.
PPT of lower Part of Sternocleidomastoid (SCM) | two minutes
  TrPs are at the lower end of this division, near its attachment to the sternum.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M. Ahmed, PHD, Study Director — University of Jazan
Locations (1):
- Jazan University, Riyadh, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data is available upon official request.